CLINICAL TRIAL: NCT04213235
Title: E.D.u.CA: a Guidebook to Increase Physical Activity Level in Cancer Patients
Brief Title: Educational Materials Development for Physical Activity in CAncer
Acronym: EDuCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alice Avancini, Investigator, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 67002
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Mixed Cancer
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical exercise (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The participants will receive the written exercise guidebook and a counselling by kinesiologist. Moreover, they will be instructed how to increase their physical activity level.

SUMMARY:
In cancer setting, physical exercise has emerged as an important factor to control cancer-related symptoms and improve patients' quality of life. In addition, the correlation between physical activity and survival is recently consolidating. Nevertheless, several previous studies have shown that the majority of cancer patients are insufficiently active. Written information, for example a guidebook, may be a good oppurtunity, to improve lifestyle. Developing and testing an exercise guidebook, based on Theory of Planned Behavior and specifically designed for cancer patients, may be an effective tool to deliver information and increase physical activity level in this population.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent;
* confirmed cancer diagnosis.

Exclusion Criteria:

- sufficient physical activity level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity level - using Godin's Leisure Time Exercise Questionnaire (GLTEQ) | Change from baseline physical activity level at 4 weeks

SECONDARY OUTCOMES:
quality of life - using European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire" (EORTC QLQ C-30) | Change from baseline physical activity level at 4 weeks
Sedentary behavior - using Sedentary Behaviour Questionnaire (SBQ) | Change from baseline physical activity level at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Italy